CLINICAL TRIAL: NCT04384588
Title: Investigational- Compassionate Use of Convalescent Plasma From COVID-19 Donors in Oncological and Non-Oncological Patients With Severity Criteria: FALP 001-2020 Trial (FALP-COVID)
Brief Title: COVID19-Convalescent Plasma for Treating Patients With Active Symptomatic COVID 19 Infection (FALP-COVID)
Acronym: FALP-COVID
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundacion Arturo Lopez Perez (Other)
Collaborators: Confederación de la Producción y del Comercio (CPC) (Unknown); Bolsa de Santiago (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FALP 001-2020
Record Dates: First submitted 2020-04-29; First posted 2020-05-12 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: COVID-19 Infection; Cancer Patients; General Population
Keywords: convalescent plasma; COVID
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Multicenter, non-randomized, 4 arms
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cancer patients with COVID 19 infection and severity criteria (Experimental): All patients will be treated with 1 or more convalescent plasma units
  Interventions: Biological: Convalescent Plasma from COVID-19 donors
- Cancer patients with COVID 19 infection and risk factors (Experimental): All patients will be treated with 1 or more convalescent plasma units
  Interventions: Biological: Convalescent Plasma from COVID-19 donors
- Non-Cancer patients COVID 19 infection and severity criteria (Experimental): All patients will be treated with 1 or more convalescent plasma units
  Interventions: Biological: Convalescent Plasma from COVID-19 donors
- Non-cancer patients COVID 19 (+) and risk factors (Experimental): All patients will be treated with 1 or more convalescent plasma units
  Interventions: Biological: Convalescent Plasma from COVID-19 donors

INTERVENTIONS:
Biological: Convalescent Plasma from COVID-19 donors — Patients that will participate in this clinical trial will be treated with Convalescent Plasma from COVID-19 donors regardless of the arm where they will be included

SUMMARY:
COVID-19 infection has spread worldwide causing several deaths in few months Convalescent Plasma from COVID 19 donors has shown huge activity in small series from Chinese patients and currently many centers from USA and the European Union are assessing its use looking to avoid mortality and prolonged hospitalizations COVID-19-related

DETAILED DESCRIPTION:
This is a collaborative, 4 arms , non randomized clinical trial assessing the use of Convalescent Plasma from COVID-19 recovered donors to be used in oncological and non-oncological patients with current severe COVID-19 infection or in patients with risk factors of major complications secondary to COVID-19 infection

ELIGIBILITY:
Inclusion Criteria:

For all patients:

A. Patient must sign an informed consent to participate in this trial

B. Signed consent to participate in this trial must be given not after 14 days from the first day of symptoms COVID-19 related

1. Patients with severity criteria must have any of the following: dyspnea and or respiratory rate >=30 per min and or saturation <= 93% with fraction of inspired oxygen 21% and or ratio of partial pressure arterial oxygen and fraction of inspired oxygen (PaFi )<300 and or lung images showing worsening in 24-48 hours

   or
2. Patients without severity criteria but with 2 or more factor risks:

A. 50 years or older

B. any of the following comorbidities: Diabetes Mellitus, Hypertension, Chronic Obstructive Pulmonary Disease, Chronic Kidney Failure, non-oncological related chronic immunosuppression

C. Total bilirubin>1,2 mg/dl or Blood Urea Nitrogen> 20 mg/dl or Lactate Dehydrogenase>245 U/L

D. D-dimer > 1mg/L

E. Neutrophils 7.3 x 10³ or greater and or Lymphocytes lesser than 0,8 x 10³ µl

F. C reactive protein >9,5 mg/dl and ferritin > 300 ug/ml

G. Interleukin-6 >7 pg/mL

H. antineoplastic treatment such as radiotherapy- cytotoxic chemotherapy- immunotherapy- molecular therapy- oncological surgery during the last 8 weeks

Exclusion Criteria:

* known allergy to plasma
* Severe multiple organic failure
* Active intra brain hemorrhage
* Disseminated intravascular coagulation with blood products requirements
* Patient with an adult respiratory distress longer than 10 days
* patients with active cancer and life expectancy shorter than 12 months according with medical criteria

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-04-07 (Actual); Primary Completion 2021-04-06 (Estimated); Study Completion 2021-04-06 (Estimated)

PRIMARY OUTCOMES:
in-hospital mortality secondary to COVID-19 among patients treated with convalescent plasma | 1 year
  in-hospital mortality secondary to COVID-19 among patients treated with convalescent plasma
safety of the use of convalescent plasma drom COVID 19 donors | 1 year
  safety of convalescent plasma from COVID 19 donors (CTCAE V5.0)

SECONDARY OUTCOMES:
Mortality at 30 days, 90 days, 6 months and 1 year | 1 year
  any cause of mortality during these periods
in-hospital Mortality COVID-19 related compared with non-treated population according to Chilean official reports | through study completion, an average of 1 year
  based on results from this trial comparing with official information
Number of days of hospitalization in high complexity facilities after convalescent plasma use | 1 year
  number of days of hospitalization in high complexity facilities after convalescent plasma use
Number of days of hospitalization in intensive care unit after convalescent plasma use | 1 year
  number of days of hospitalization in intensive care unit after convalescent plasma use
Number of days of mechanical ventilatory support in patients after convalescent plasma use | 1 year
  number of days of mechanical ventilatory support in patients after convalescent plasma use
Total number of days of mechanical ventilatory support | 1 year
  total number of days of mechanical ventilatory support
Total number of hospitalization days in patients treated with convalescent plasma | 1 year
  total number of hospitalization days in patients treated with convalescent plasma
Number of hospitalization days in patients after treatment with convalescent plasma | 1 year
  total number of hospitalization days in patients after treatment with convalescent plasma
Viral load measuring | 14 days
  Viral load measuring
Immunological response in treated patients (COVID19-Immunoglobulin M and Immunoglobulin G, neutralizing antibodies) | day 1 of hospitalization
  COVID19-Immunoglobulin M and Immunoglobulin G, neutralizing antibodies
Negativization of COVID 19 load since convalescent plasma use | 14 days
  negativization of COVID 19 load since convalescent plasma use
Negativization of COVID 19 load since hospitalization | 14 days
  negativization of COVID 19 load since hospitalization
Negativization of COVID 19 load since first reported symptoms COVID-19 related | 14 days
  negativization of COVID 19 load since first reported symptoms COVID-19 related
Donor Interferon Gamma profile characterization | 1 day
  Interferon Gamma measurement from donor
Donor Granulocyte Macrophage Colony Stimulating Factor characterization | 1 day
  Granulocyte Macrophage Colony Stimulating Factor measurement from donor
Donor Tumor Necrosis Factor Alfa characterization | 1 day
  Tumor Necrosis Factor Alfa measurement from donor
Donor Interleukin -1 beta characterization | 1 day
  Interleukin -1 beta measurement from donor
Donor Interleukin-2 characterization | 1 day
  Interleukin -2 measurement from donor
Donor Interleukin-4 characterization | 1 day
  Interleukin -4 measurement from donor
Donor Interleukin-6 characterization | 1 day
  Interleukin -6 measurement from donor
Donor Interleukin-8 characterization | 1 day
  Interleukin -8 measurement from donor
Donor Interleukin-10 characterization | 1 day
  Interleukin -10 measurement from donor
Receptor Interferon Gamma profile characterization | 1 day
  Interferon Gamma measurement from receptor
Receptor Granulocyte Macrophage Colony Stimulating Factor characterization | 1 day
  Granulocyte Macrophage Colony Stimulating Factor measurement from receptor
receptor Tumor Necrosis Factor Alfa characterization | 1 day
  Tumor Necrosis Factor Alfa measurement from receptor
receptor Interleukin -1 beta characterization | 1 day
  Interleukin -1 beta measurement from receptor
Receptor Interleukin-2 characterization | 1 day
  Interleukin -2 measurement from receptor
Receptor Interleukin-4 characterization | 1 day
  Interleukin -4 measurement from receptor
Receptor Interleukin-6 characterization | 1 day
  Interleukin -6 measurement from receptor
Receptor Interleukin-8 characterization | 1 day
  Interleukin -8 measurement from receptor
Receptor Interleukin-10 characterization | 1 day
  Interleukin -10 measurement from receptor

CONTACTS AND LOCATIONS:
Overall Officials: Raimundo Gazitua, MD, Principal Investigator — Fundacion Arturo Lopez Perez
Locations (1):
- Fundacion Arturo Lopez Perez, Providencia, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No